CLINICAL TRIAL: NCT04521283
Title: Visual Outcome of Traumatic Posterior Segment Complications in Upper Egypt :Tertiary Center Study
Brief Title: Visual Outcome of Traumatic Posterior Segment Complications
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Rehab Azzam, Principle investigator, Assiut University
Other Study IDs: traumatic posterior segment
Record Dates: First submitted 2020-08-18; First posted 2020-08-20 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Eye Injuries
MeSH Terms: conditions — Eye Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
to identify the demographic, the clinical characteristics and the possible predictive factors affecting long-term visual outcomes of traumatic posterior segment complications presenting to Assiut University Hospital.

DETAILED DESCRIPTION:
Ocular trauma is an important public health problem which is preventable and its etiology, severity, and outcome depends on many factors in the changing environment . Even eyes represent only 0.27% of the body surface area and 4% of the facial area, they are the third most commonly trauma-exposed area after the hands and feet . It is estimated that, worldwide, there are approximately 1.6 million people blind from eye injuries, 2.3 million bilaterally visually impaired and 19 million with unilateral visual loss; these facts make ocular trauma the most common cause of unilateral blindness . In population-based surveys, the percentage of monocular blindness due to trauma ranged from 20% to 50% and of bilateral blindness from 3.2% to 5.5% .

Ocular injuries vary with a broad range of severity and include simple subconjunctival injury, lid laceration, corneal abrasion, traumatic iritis, hyphaema, lens injury, vitreous haemorrhage (VH) , retinal detachment, traumatic optic neuropathy, retrobulbar haemorrhage, orbital fracture, and ruptured globes. Ocular injuries are classified into 2 groups as open and close globe injuries. Ruptured globes fall into the category of open globe injuries, which are injuries resulting in a full-thickness laceration of the cornea and/or sclera. Wounds can be penetrating (with one entry wound and no exit wound), or perforating (a through-and-through injury with both entrance and exit wounds) . Closed globe injuries resulting from blunt trauma can cause hyphaema, vitreous haemorrhage, retinal tears and detachment, choroidal rupture, macular oedema, and even globe rupture, retrobulbar haemorrhage and traumatic optic neuropathy .

In Kasr El Aini Hospital The majority of ocular trauma in their population was due to assaultive injuries occurring mainly in males. Open globe injuries were more common than closed globe injuries, and globe lacerations were more common than ruptured globes .

IN Upper Egypt Pediatric ocular trauma among patients referred to their tertiary ophthalmology referral center over a period of 1 year was 3.7%. Of these, 67.3% of cases had open globe injury, 30.7% had closed injury, and only 2% had chemical injury.

Posterior segment ocular trauma is still an important cause of visual loss and disability in working-age population. With modern surgical approaches, many eyes can be salvaged with retention of vision(9). These complications are retinal detachment (RD), vitreous hemorrhage(VH), posterior intraocular foreign body (IOFB), dislo-cated lens, choroidal detachment(10)

ELIGIBILITY:
Inclusion Criteria:

All patients presenting with traumatic posterior segment complications in outpatient clinics and operative rooms

Exclusion Criteria:

* A history of recent intraocular surgery
* No history of trauma.
* Loss to follow-up

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who underwent traumatic posterior segment complications of the eye
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2021-08-01 (Estimated); Study Completion 2021-08-01 (Estimated)

PRIMARY OUTCOMES:
Visual outcome of traumatic vitreous haemorrhage | One year
  • The initial and final visual acuity outcomes will be compared to identify subjects who witnessed any improvement in their visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Samir Y Salah, Professor, Study Director — Assiut University; Abdelsalam Abdallah, Professor, Study Director — Assiut University; Dalia M Eltohamy, Lecturer, Study Director — Assiut University